CLINICAL TRIAL: NCT00996450
Title: Educational Follow-up in a Cohort of Children at the Royal Marsden Hospital, Following the Treatment of a Brain Tumour
Brief Title: Educational Follow-up in a Cohort of Children at the Royal Marsden Hospital (RMH)
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR2903
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2009-10

CONDITIONS: Brain Tumour
Keywords: brain tumour
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To document pre-diagnosis educational abilities, to document any change in educational achievements following treatment, to document educational support given within the statement process and to document the timing of support.

DETAILED DESCRIPTION:
This will be a retrospective study. Cases will be identified by looking at the Royal Marsden Hospital (RMH) coding database. All the patients will have completed treatment for a brain tumour. The children all need to have started school before the diagnosis of their brain tumour so that we can look at easily defined educational assessments in this cohort. Children will be identified by looking at RMH coding of diagnosis and include children aged between 4 years and 18 years old (school age).

ELIGIBILITY:
Inclusion Criteria:

* patients/parental consent for RMH accessing educational information from them and their school
* patients with a primary brain tumour

Exclusion Criteria:

* children with secondary brain tumours
* children who have had treatment for a relapse of primary brain tumour

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cases will be identified by looking at RMH coding database. Medical information will be sort from the electronic patient records (EPR) and from the patient notes.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

SECONDARY OUTCOMES:
To compare educational achievements of children of different tumour types following treatment.
To document if there are any differences in educational achievements depending on the age at diagnosis of the brain tumour.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Darren Hargrave, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Belmont, Surrey, United Kingdom